CLINICAL TRIAL: NCT04651595
Title: Efficacy of Caudal Block on Intra-operative Anal Sphincter Muscle Tone and Post-operative Analgesia During Anal Sphincter Sparing Procedures Under General Anaesthesia: A Randomized Control Trial
Brief Title: Efficacy of Caudal Block on Intra-operative Anal Sphincter Muscle Tone and Post-operative Analgesia During Anal Sphincter Sparing Procedures Under General Anaesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, Ayman Abougabal, lecturer of anaesthesia, SICU and pain management, Kasr El Aini Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: N-33-2019
Record Dates: First submitted 2020-11-26; First posted 2020-12-03 (Actual); Last update posted 2022-10-20 (Actual); Status verified 2022-10

CONDITIONS: Efficacy of Caudal Block on Intra-operative Anal Sphincter Muscle Tone
MeSH Terms: interventions — Morphine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Caudal (Experimental)
  Interventions: Procedure: Caudal block
- Control (Active Comparator)
  Interventions: Drug: Morphine

INTERVENTIONS:
Procedure: Caudal block — caudal block with low dose bupivicaine 0.25% to preserve tone
  Arms: Caudal
Drug: Morphine — morphine to control pain and avoid using muscle relaxant
  Arms: Control

SUMMARY:
upplementing general anaesthesia with caudal analgesia in sphincter sparing procedures might be useful as it will provide a satisfactory combination of sphincter muscle tone preservation, good intraoperative and postoperative analgesia along with a reduction in the consumption of opioids and anaesthetic drugs. To the best of our knowledge, this anaesthetic technique was not tested in sphincter sparing procedures before.

DETAILED DESCRIPTION:
Anal fistulae, defined as an abnormal connection between the distal alimentary tract and the integument, are among the common illnesses affecting the anal canal, with a prevalence rate of 8.6 cases per 100,000.1 Usually, anorectal fistulae are safely and reliably treated by fistulotomy. One of the common complications of fistulotomy is incontinence due to sphincter injury, with an incidence reaching up to 12%2. Moreover, this technique is not well suited for complex anal fistulae due to the prevalent risk of incontinence reaching up to 50%2. That created the need for sphincter sparing procedures to evolve which do not involve division of any portion of the sphincter complex, thus evolvement of an anaesthetic technique which spares the presence of muscle tone, and provides good postoperative analgesia.2,3 The choice of anaesthetic technique for sphincter sparing procedures is challenging. Regional anaesthetic techniques such as saddle, lumbar epidural, and caudal blocks are considered well tolerable and reliable for anorectal surgery. Lumbar epidural local anaesthesia does not produce a uniform anaesthetic effect across the spinal segments as the large size of the L5 and S1 nerve roots may be resistant to the local anaesthetic effect and The cranial spread of lumbar epidural anaesthesia is somewhat more extensive than the caudal spread which suggest that the onset of the block of the caudal sacral segments may be later than that of the lumbar segments. 4On the other hand, saddle anaesthesia is the preferred route for most of the anorectal surgeries as it abolishes the muscle tone5; however, loss of the muscle tone consequently increases the possibility of the external anal sphincter injury in complex anal fistulas. Thus; sphincter sparing procedures are usually performed under general anaesthesia omitting neuromuscular blocking agents in order to preserve sphincter tone intraoperatively.6 However, the choice of general anaesthesia for this procedure still lacks adequate postoperative analgesic plan.

Caudal block is not a commonly used route for analgesia in adults due to the evolution of lumbar epidural block5. The introduction of ultrasound for guiding different blocks, including caudal block had increased the use of caudal block7 especially when sacral nerve spread of anaesthetics is preferred over lumbar nerve spread8. Modern epidural dosing regimens (e.g. 0.0625% to 0.1 % bupivacaine with 2-4 mcg/ml fentanyl) 6,9 reduce the total local anaesthetic dose required and motor block experienced; potentially allowing the patient to be ambulatory.

Therefore, Supplementing general anaesthesia with caudal analgesia in sphincter sparing procedures might be useful as it will provide a satisfactory combination of sphincter muscle tone preservation, good intraoperative and postoperative analgesia along with a reduction in the consumption of opioids and anaesthetic drugs. To the best of our knowledge, this anaesthetic technique was not tested in sphincter sparing procedures before.

ELIGIBILITY:
Inclusion Criteria:

- with complex anal fistula -

Exclusion Criteria:

* known hypersensitivity to amide type local anesthetics, contraindications to caudal block such as use of anticoagulant medication, local infection in the intervention site, increased intracranial pressure, severe aortic and / or mitral valve stenosis, and ischemic hypertrophic sub aortic stenosis, along with BMI (Body mass index) > 35 kg/m2 , anatomical abnormalities or previous surgeries involving the sacrum.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
The time to first request of rescue postoperative analgesic | in the first 24 hour
  the time interval between the end of surgery and the first request to postoperative morphine

SECONDARY OUTCOMES:
Digital Rectal Examination Scoring System (DRESS | intraoperative
  Digital Rectal Examination Scoring System to asses the anal tone

CONTACTS AND LOCATIONS:
Locations (1):
- Kasr alainy medical school, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided